CLINICAL TRIAL: NCT00391729
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Dose-Ranging Study of the Safety and Efficacy of ABT-089 in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: A Dose-Ranging, Cross-over Study of the Safety and Efficacy of ABT-089 in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M06-855
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — pozanicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: ABT-089

INTERVENTIONS:
Drug: ABT-089 — Subjects will take 2 mg QD, 5 mg QD, 15 mg QD, 40 mg QD, 40 mg BID for 4-6 weeks
  Arms: 2
Drug: Placebo — Subjects will take placebo QD, BID for 4-6 weeks
  Arms: 1

SUMMARY:
The objective of this study is to compare the safety and efficacy of five doses of ABT-089 (2 mg QD, 5 mg QD, 15 mg QD, 40 mg QD and 40 mg BID) to placebo in adults with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for attention deficit hyperactivity disorder
* Have voluntarily signed an informed consent form
* Are between 18 and 60 years of age
* Will use contraceptive methods during the study
* Women must not be pregnant or breast-feeding
* Must be in generally good health
* Are fluent in English

Exclusion Criteria:

* They have a current or past diagnosis of schizoaffective disorder, schizophrenia, obsessive-compulsive disorder, drug-induced psychosis, bipolar disorder, psychotic disorder or mental retardation
* They have a current diagnosis of major depressive episode, generalized anxiety disorder (GAD), or post-traumatic stress disorder (PTSD) or have a clinically significant sleep disorder requiring treatment
* They require ongoing treatment or expected treatment with any psychotropic medication, including anxiolytics, antipsychotics, anticonvulsants, antidepressants or mood stabilizers
* They failed to respond to two or more adequate trials of FDA-approved ADHD medication
* They have violent, homicidal or suicidal ideation
* They have a significant history of medical diagnoses, seizure disorder, Tourette's syndrome or a central nervous system (CNS) disease, excluding ADHD
* They have a urine drug screen that is positive for alcohol or drugs of abuse
* They have a history of substance or alcohol disorder (abuse/dependence) during the last 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Investigator-rated Connors' Adult ADHD Rating Scale(CAARS) total score | at the final evaluation of each 4-week treatment period

SECONDARY OUTCOMES:
CAARS Inattentive and Hyperactive/Impulsive Sub scales Scores | at the final evaluation of each 4-week treatment period
CAARS ADHD Index, CAARS:Self | at the final evaluation of each 4-week treatment period
CGI-ADHD-S, AISRS, TASS, FTND | at the final evaluation of each 4-week treatment period
QSU-Brief, CANTAB cognitive battery | at the final evaluation of each 4-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gault, MD,PhD, Study Director — Abbott
Locations (23):
- United States (23):
  - Mesa, Arizona
  - Lafayette, California
  - Oceanside, California
  - San Diego, California
  - Denver, Colorado
  - Jacksonville, Florida
  - Maitland, Florida
  - Miami, Florida
  - Tampa, Florida
  - Newton, Kansas
  - Farmington Hills, Michigan
  - Omaha, Nebraska
  - Bridgewater, New Jersey
  - New York, New York
  - Staten Island, New York
  - Chapel Hill, North Carolina
  - Lyndhurst, Ohio
  - Portland, Oregon
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Lake Jackson, Texas
  - Herndon, Virginia
  - Middleton, Wisconsin

REFERENCES:
- [Derived] Apostol G, Abi-Saab W, Kratochvil CJ, Adler LA, Robieson WZ, Gault LM, Pritchett YL, Feifel D, Collins MA, Saltarelli MD. Efficacy and safety of the novel alpha(4)beta(2) neuronal nicotinic receptor partial agonist ABT-089 in adults with attention-deficit/hyperactivity disorder: a randomized, double-blind, placebo-controlled crossover study. Psychopharmacology (Berl). 2012 Feb;219(3):715-25. doi: 10.1007/s00213-011-2393-2. Epub 2011 Jul 12. PMID 21748252